CLINICAL TRIAL: NCT07002489
Title: A Single-arm, Open-label Study of Efficacy of Notrande Shuhuajun Probiotic Supplement on Lmproving Constipation in Preschool Children Aged 3-6
Brief Title: Efficacy of Notrande Shuhuajun Probiotic Supplement on Lmproving Constipation in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Sibote Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-RD-04-JJ-001
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Functional Constipation (FC)
Keywords: probiotics; constipation; functional constipation; pre-school children
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Notrande Shuhuajun Probiotic Supplement Study Product (Other): Notrande Shuhuajun Probiotic Supplement, Each capsule contains the following active ingredients: ≥79.5 mg of the specially developed formula, 1 × 108 CFU of Lactobacillus fermentum CECT5716, 5 × 109 CFU of Lactobacillus rhamnosus GG, 5 × 109 CFU of Bifidobacterium animalis (Lactobacillus subspecies HNO19), and 1 × 108 CFU of Lactobacillus rhamnosus HNO01.
  Interventions: Dietary Supplement: Nuotelande Shuhuajun Study Product

INTERVENTIONS:
Dietary Supplement: Nuotelande Shuhuajun Study Product — Participants in this arm need to take in the assigned product - Notrande Shuhuajun Probiotic Supplement, 1 capsule per day, for 14 consecutive days. Don't take in similar products in the following 7 days (regression phase).

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of Notrande Shuhuajun Probiotic Supplement intake on the improvement of functional constipation in preschool children (3-6 years old). The main questions it aims to answer are:

- Does Notrande Shuhuajun Probiotic Supplement intake improve functional constipation in preschool children?

105 eligible participants will be enrolled in one center and assigned the study product. After one week washout period participants need to take in the product for two weeks, followed by a one-week regression period.

Researchers will collect data, analyze data and conclude whether the study product is effective to improve constipation in participants, by comparing the change of concentration of biochemical indicators SCFA (Short-chain fatty acids), Lactobacillus and Bifidobacterium, and visual analysis of Bristol Stool scale etc..

ELIGIBILITY:
Inclusion Criteria:

* Participants must be preschool children (aged 3-6);
* Participants were diagnosed with functional constipation based on Rome IV criteria;
* Participants agreed not to take any drugs, supplements, or other dairy products during the trial period;
* Participants agreed not to take any other prebiotic/bacterial drugs, supplements, or dairy products including yogurt beverages during the trial period;
* Be willing to refrain from participating in other interventional clinical studies during the trial period;
* Be able to fully understand the nature, purpose, benefits obtained, as well as possible risks and side effects of this study;
* Be willing to comply with all test requirements and procedures;
* Sign the informed consent form;

Exclusion Criteria:

* In the treatment of gastrointestinal symptoms;
* Lactose intolerance;
* Currently suffering from other organic diseases that affect intestinal function, such as a history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, congenital megacolon, scleroderma, anorexia nervosa, etc;
* Have been controlling diet, increasing exercise, or taking drugs to control weight or affect appetite in the last three months;
* Have any of the following medical histories or have been clinically diagnosed with any of the following diseases that may affect the evaluation of the trial effect: obvious gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases;
* Current or past abuse of alcohol or other prohibited drugs, supplements or OTC prescription drugs may cause intestinal dysfunction or affect the evaluation of the test results;
* According to the researchers' judgment, drugs that may affect gastrointestinal function or the immune system are currently being frequently used;
* Laxatives or other digestive AIDS were used two weeks before the start of the trial;
* Have consumed dairy products or other foods containing prebiotics/bacteria 10 days before the start of the trial;
* The research doctors believed that the volunteers could not fully cooperate with the trial arrangements;

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-24 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Change of constipation indicators-SCFA (Short-chain fatty acids) level in the fecal samples | day 0, day 14, and day 21
  Change of constipation indicators: SCFA (Short-chain fatty acids) level in the fecal samples, from baseline day 0, to day 14, and to end day 21. unit: mg/100g fecal sample, higher level means improved constipation.
Change of constipation indicators- Probiotics - Lactobacillus and Bifidobacterium concentration level in the fecal samples | day 0, day 14, and day 21
  Change of constipation indicators: Probiotics - Lactobacillus and Bifidobacterium concentration level via qPCR in the fecal samples, from baseline day 0, to day 14, and to end day 21. unit: CFU/g, higher level means improved constipation.

SECONDARY OUTCOMES:
Change of Bristol Stool Form Scale (BSFS) | day 0 , day 21
  Change of Bristol Stool Form Scale (BSFS) by visual judgement of look and form of participants' bowel movements, type 1 to type 7, mapping to score 1 to 7, the smaller value indicates improved constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — Raison Biotech Group
Locations (1):
- Fuyang Fifth People's Hospital Quanying Branch, Fuyang, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
The abstract of final clinical study report will be shared via official website.
Supporting Information: CSR
Time Frame: The abstract of final clinical study report is available since Dec 15, 2025, and will last until otherwise notified.
Access Criteria: Any one can access, and the public link will be shared once available
URL: http://www.raisonbiotech.com/Data/25-RD-04-JJ-001-Abstract-ENv4.pdf